CLINICAL TRIAL: NCT02041338
Title: Phase 2 Randomized Study of Different Neoadjuvant Regimens in Subtypes of Breast Cancer
Brief Title: Study of Optimizing Neoadjuvant Regimens in Subtypes of Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Binghe Xu, MD, professor and Director of Department of Medical Oncology, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-BC-026
Record Dates: First submitted 2014-01-15; First posted 2014-01-22 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-02

CONDITIONS: Breast Cancer; Neoadjuvant Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Carboplatin; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Luminal subtype test (Experimental): Paclitaxel 175mg/m2, every 2 weeks as a cycle for 4-6 cycles
  Interventions: Drug: Paclitaxel
- Luminal subtype control (Active Comparator): Epirubicin 75mg/m2 plus paclitaxel 175mg/m2 every 3 weeks as a cycle for 4-6 cycles
  Interventions: Drug: Epirubicin and Paclitaxel
- Her2 positive subtype test (Experimental): Paclitaxel 175mg/m2 plus carboplatin AUC 4 with or without trastuzumab every 2 weeks as a cycle for 4-6 cycles
  Interventions: Drug: Paclitaxel and carboplatin
- Her2 positive subtype control (Active Comparator): Epirubicin 75mg/m2 plus paclitaxel 175mg/m2 with or without trastuzumab every 3 weeks as a cycle for 4-6 cycles
  Interventions: Drug: Epirubicin and Paclitaxel
- Triple negative subtype test (Experimental): Paclitaxel 175mg/m2 plus carboplatin AUC 4 every 2 weeks as a cycle for 4-6 cycles
  Interventions: Drug: Paclitaxel and carboplatin
- Triple negative subypte control (Active Comparator): Epirubicin 75mg/m2 plus paclitaxel 175mg/m2 every 3 weeks as a cycle for 4-6 cycles
  Interventions: Drug: Epirubicin and Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel and carboplatin
  Arms: Her2 positive subtype test; Triple negative subtype test
Drug: Paclitaxel
  Arms: Luminal subtype test
Drug: Epirubicin and Paclitaxel
  Arms: Her2 positive subtype control; Luminal subtype control; Triple negative subypte control

SUMMARY:
There are no standard neodjuvant regimens adapted according to the different subtypes of breast cancer. This is a phase 2, randomized study to evaluate several regimens in different subtypes of breast cancer.

DETAILED DESCRIPTION:
Breast cancer is a heterogenous disease with at least 4 intrinsic subtypes including Luminal A, Luminal B, HER2 enriched, Basal-like and normal breast like. Different subtypes have different prognosis and treatment sensitivity. Thus, it would be more suitable to administer different chemo-regimen in different subtypes. This is especially true in neoadjuvant chemotherapy setting where no standard regimen has ever been established. Therefore, we designed this phase 2 randomized clinical trial to explore potential effective regimens in variable subtypes of breast cancer in neoadjuvant treatment. Patients were first classified into Luminal type, Her2 positive type and triple-negative type by immunohistochemistry exam of ER/PR/HER2 in core needle biopsy and then randomized to received either dose dense paclitaxel in Luminal type or dose dense paclitaxel plus carboplatin with or without trastuzumab in HER2 positive type or dose dense paclitaxel plus carboplatin in triple-negative type.The control groups in each subtype all receive paclitaxel plus epirubicin every 3 weeks. The duration of treatment is 4-6 cycles. Primary endpoint is the pathological CR rate in each subtypes. Secondary endpoints include disease free survival, objective response rate, safety. Tissue samples and blood samples will be collected at baseline and during treatment. There will be exploratory biomarkers analyses to identify predictive markers for efficacy in every subtypes.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIa-IIIc breast cancer patients plan to receive neoadjuvant chemotherapy
* Patients have enough tissue sample to do IHC test for subtype classification
* Patients have at least one measurable lesion according to RECIST1.1
* KPS≥80
* No prior treatment for breast cancer
* Adequate bone marrow (neutrophil count ≥1500 ml and platelet count ≥100,000 ml), renal (serum creatinine <1.5 times the upper limit of normal [ULN] or a creatinine clearance of ≥60 ml/minute), hepatic (total bilirubin ≤1.5 ULN; alanine aminotransferase, aspartate aminotransferase, and alkaline phosphatase ≤2.5 ULN), and cardiac function (assessed by electrocardiogram or thoracic radiography) were required.

Exclusion Criteria:

* Fertile women were excluded if pregnant or lactating or if they were not using adequate contraception.
* Previous chemotherapy for breast cancer.
* history of other serious illness (e.g. congestive heart failure, angina pectoris, uncontrolled hypertension or arrhythmia, clinically significant neurologic or psychiatric disorders, uncontrolled serious infection, AIDS), had an organ allograft, severe gastrointestinal disorder, or other neoplasias (except for in situ cervical cancer, non-melanoma skin cancer, or previous diagnosis of cancer with no evidence of disease for >10 years).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
pathological complete response(pCR) rate of breast and axilla after surgery | 3 years
  pathological complete response(pCR) of breast and axilla after surgery means after operation, no invasive component can be found in both breast and axillary lymph nodes. The pCR rate is calculated by number of patients having pCR after sugery divided by number of patients receiving neoadjuvant chemotherapy.

SECONDARY OUTCOMES:
Disease free survival | 3years and 5years after operation
Overall survival | 3 years and 5years after operation
Adverse event | during screening and treatment, withing 21 days after day 1 of last cycle

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China